CLINICAL TRIAL: NCT02906787
Title: Behavioral Activation for Smoking Cessation and the Prevention of Post-Cessation Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 825425; R01CA206058 (NIH); NCT03254433 (obsolete NCT alias)
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Results first posted 2023-02-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Smoking Cessation; Weight Loss
Keywords: Smoking Cessation; Weight Loss
MeSH Terms: conditions — Smoking Cessation; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAS+ (Experimental): Participants will attend 8 counseling sessions and receive a behavioral activation intervention to smoking cessation and to post-cessation weight gain (BAS+).
  Interventions: Behavioral: BAS+
- SC (Placebo Comparator): Participants will attend 8 counseling sessions and receive standard smoking cessation counseling (SC).
  Interventions: Behavioral: SC

INTERVENTIONS:
Behavioral: BAS+ — The goal of the BAS+ is to maintain a level of overall reward after cessation by structuring and enhancing opportunities for reinforcement to: (1) ensure that not smoking is as reinforcing as smoking; and (2) prevent an over-reliance on food as a substitute reinforcer for smoking so that PCWG does not precipitate smoking relapse.
  Arms: BAS+
Behavioral: SC — Overeating and weight gain are common concerns reported during smoking cessation treatment. Per convention, SC will address these concerns through standard recommendations to consume low-calorie snack foods, drink water, eat nutritious meals, and exercise, but will not include skills to shape the use of these suggestions.
  Arms: SC

SUMMARY:
The purpose of this research study is to better understand (1) why people gain weight when they quit smoking and (2) whether certain types of smoking cessation (i.e. quit smoking) counseling combined with the nicotine patch help people quit smoking and gain less weight.

DETAILED DESCRIPTION:
This is a randomized clinical trial of the efficacy of a behavioral activation intervention to smoking cessation and to post-cessation weight gain (BAS+) plus transdermal nicotine (TN) compared to standard smoking cessation counseling (SC) plus TN in treatment-seeking smokers. After completing an Intake Visit (~week -3), eligible smokers will be randomized (stratified by nicotine dependence, BMI and gender) to participate in 8 individual sessions of BAS+ or SC over a 10-week treatment period with two sessions prior to the target quit date (weeks -2, -1) and six sessions post-target quit date (TQD [week 0] and weeks 1, 2, 4, 6, and 8). Standard, 8-week; open-label TN will begin on the TQD. Moderators will be assessed pre-treatment. Mediating mechanisms will be assessed before, during, and at the end of treatment (EOT, week 8). Smoking will be assessed by self-report and biochemically confirmed (Carbon Monoxide [CO] < 5) at all in-center visits after quitting, at EOT (week 8), and at the 12- and 26-week follow-ups. Weight will be assessed at these same time points. Food intake will be measured by three consecutive days of 24-hour food recalls at Baseline [week -2] and 4-, 8-, and 12- and 26-weeks post-TQD. Smoking cessation and post-cessation weight gain (PCWG) are the primary outcomes and food intake is a secondary outcome at 26-weeks post-TQD. Consistent with intent-to-treat (ITT) analyses, the investigators will measure smoking cessation and weight gain in the full sample at the 26-week follow-up, evaluating a smoking status by treatment interaction for the PCWG analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female treatment-seeking smokers who are between 18 and 65 years of age and self-report smoking at least 5 cigarettes (menthol and/or non-menthol) per day for at least the last 6 months.
* Plan to live in the area for the duration of the study (i.e. ~30 weeks/8 months).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
* Smokers who wish to make a permanent quit attempt in the next 1-2 months (treatment-seeking), because our prior work suggests that motivated subjects are more sensitive to medication effects on smoking behavior.
* Able to communicate fluently in English (i.e. speaking, writing, and reading).
* Provide a Carbon Monoxide (CO) breath test reading greater than or equal to 5 parts per million (ppm) at the Intake Visit.

Exclusion Criteria:

Smoking Behavior.

* Regular use of nicotine containing products other than cigarettes (e.g. chewing tobacco, snuff, snus, cigars, e-cigs, etc.). Participants agreeing to abstain from using nicotine containing products other than cigarettes and the study-provided TN for the duration of trial will be considered eligible.
* Current enrollment or plans to enroll in another research and/or smoking cessation program over the duration of the study (i.e. ~30 weeks/8 months).
* Anticipated use (within the next ~30 weeks/8 months) of any nicotine substitutes and/or smoking cessation treatments/medications unless provided through the study.
* Provide a CO breath test reading less than 8 ppm at Intake Visit.

Alcohol and Drug.

* History of substance abuse (other than nicotine) in the past 12 months and/or currently receiving medical treatment for substance abuse. Counseling and support groups (e.g. Alcoholics Anonymous and Narcotics Anonymous) will not be considered medical treatment for the purposes of this protocol.
* Current alcohol consumption that exceeds 25 standard drinks/week.
* Breath alcohol reading (BrAC) greater than .000 at the Intake Visit.
* A positive urine drug screen (UDS) for cocaine, opiates, amphetamines, methamphetamines, phencyclidine (PCP), ecstasy (MDMA), barbiturates, benzodiazepines, methadone, and/or oxycodone at the Intake Visit.

Medical.

* Women who are pregnant, breast feeding, or planning a pregnancy over the duration of the study period. Women must agree to use an adequate form of contraception or abstain from sexual intercourse for the duration and for at least one month after the end of the study.
* Current treatment of cancer or diagnosed with cancer (except basal or squamous-cell carcinoma not treated with chemotherapy and/or radiation) in the past 6 months.
* Poorly controlled, brittle, or pump-dependent Type I diabetes.
* Current peptic ulcer bleeding.
* Allergy to adhesive tape.
* Skin problems or sensitivities. Eligibility will be evaluated on a case-by-case basis by the Study Physician.
* Active hepatitis or poorly controlled kidney and/or liver disease.
* Uncontrolled hypertension (systolic blood pressure [SBP] greater than 159 and/or diastolic blood pressure [DBP] greater than 99
* History of abnormal heart rhythms, tachycardia, and/or cardiovascular disease (e.g. stroke, angina, heart attack) may result in ineligibility. These conditions will be evaluated on a case-by-case basis by the Study Physician.
* History of epilepsy or seizures. Eligibility will be evaluated on a case-by-case basis by the Study Physician.
* Serious or unstable disease within the past 6 months. Notable diseases will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Any impairment including, but not limited to, visual, physical, and/or neurological impairments preventing proper completion of the study procedures. Notable impairments will be evaluated on a case-by-case basis by the Principal Investigator and/or the Study Physician.
* Low or borderline intellectual functioning - determined by receiving a score of less than 75 on the Shipley Institute of Living Scale (SILS), which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated Intelligence Quotient (IQ) Test.
* Applicable food allergies or disorders:

Galactosemia, Notable milk allergy (lactose intolerant participants may proceed unless they experience severe symptoms), Notable soy allergy, Peanut allergy

Psychiatric.

* Current diagnosis of major depression. Subjects with a history of major depression, in remission for 6 months or longer (may be stable on antidepressant medications), are eligible.
* Lifetime history of a suicide attempt.
* Lifetime history of schizophrenia, psychosis, and/or bipolar disorder.

Medication.

Current use or recent discontinuation (within the last 14 days) of:

* Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin Standard-Release, Chantix).
* Anti-psychotic medications.
* Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
* Systemic steroids.

Current use of:

* Nicotine replacement therapy (NRT).
* Heart medications such as digoxin, quinidine, and nitroglycerin.

Daily use of:

* Opiate-containing medications for chronic pain.
* Inhaled corticosteroids.
* Benzodiazepines and/or Barbiturates.

General Exclusion.

* Past, current, anticipated, or pending enrollment in another research program over the study period that could potentially impact subject safety, study data, and/or the study design as determined by the Principal Investigator and/or Study Physician.
* Any medical condition, illness, disorder, adverse event (AE), or concomitant medication that could compromise participant safety or significantly impact study performance as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible for any of the aforementioned reasons at any point throughout the study, as well as during the initial telephone screen.
* Significant non-compliance with protocol and/or study design as determined by the Principal Investigator and/or Study Physician. Subjects may be deemed ineligible at any point throughout the study.
* Subjects failing to complete an in-person Baseline Visit will be excluded (no Principal Investigator determination required).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Audrain-McGovern, Ph.D., Principal Investigator — Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Audrain-McGovern J, Wileyto EP, Ashare R, Albelda B, Manikandan D, Perkins KA. Behavioral activation for smoking cessation and the prevention of smoking cessation-related weight gain: A randomized trial. Drug Alcohol Depend. 2023 Mar 1;244:109792. doi: 10.1016/j.drugalcdep.2023.109792. Epub 2023 Feb 1. PMID 36739753

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard SC: Participants will attend 8 counseling sessions and receive standard smoking cessation counseling (SC).
  SC: Overeating and weight gain are common concerns reported during smoking cessation treatment. Per convention, SC will address these concerns through standard recommendations to consume low-calorie snack foods, drink water, eat nutritious meals, and exercise, but will not include skills to shape the use of these suggestions.
Period: Overall Study
Arm/Group | BAS+ | Standard SC
Started | 142 | 146
EOT | 106 | 112
3-month Follow-up | 106 | 114
Enrolled in Neuroimaging Sub-study | 31 | 28
Neuroimaging Sub-study: Completed Scan 1 | 30 | 26
Neuroimaging Sub-study: Completed Scan 2 | 25 | 20
Neuroimaging Sub-study: Completed EOT | 25 | 20
Neuroimaging Sub-study: Completed 12-Week Follow-up | 25 | 20
Completed Neuroimaging Sub-study | 25 | 20
Completed | 106 | 114
Not Completed | 36 | 32
Not completed — Withdrawal by Subject | 12 | 10
Not completed — Missed | 24 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BAS+ | Standard SC | Total
Number analyzed (Participants) | 142 | 146 | 288
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  years
    Main Study Participants | 46.01 (12.30) | 45.97 (12.01) | 45.99 (12.13)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 45.56 (12.66) | 42.32 (10.49) | 44.11 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  Participants
    Main Study Participants: Female | 57 | 62 | 119
    Main Study Participants: Male | 85 | 84 | 169
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants: Female | 10 | 7 | 17
    Sub-Study Participants: Male | 15 | 12 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  Participants
    Main Study Participants: Black/African American | 85 | 86 | 171
    Main Study Participants: White | 51 | 50 | 101
    Main Study Participants: Unknown or not reported | 6 | 10 | 16
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants: Black/African American | 11 | 8 | 19
    Sub-Study Participants: White | 14 | 8 | 22
    Sub-Study Participants: Unknown or not reported | 0 | 3 | 3
Education [Count of Participants; unit: Participants] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  Participants
    Main Study Participants: HS Graduate or less | 51 | 54 | 105
    Main Study Participants: Some College | 55 | 54 | 109
    Main Study Participants: College Graduate | 36 | 38 | 74
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants: HS Graduate or less | 8 | 4 | 12
    Sub-Study Participants: Some College | 6 | 10 | 16
    Sub-Study Participants: College Graduate | 11 | 5 | 16
Income [Count of Participants; unit: Participants] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  Participants
    Main Study Participants: < $20,000 | 54 | 45 | 99
    Main Study Participants: $20,000 - $50,000 | 57 | 73 | 130
    Main Study Participants: > $50,000 | 31 | 28 | 59
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants: < $20,000 | 8 | 8 | 16
    Sub-Study Participants: $20,000 - $50,000 | 8 | 6 | 14
    Sub-Study Participants: > $50,000 | 9 | 5 | 14
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  cigarettes per day
    Main Study Participants | 14.18 (6.36) | 14.33 (7.61) | 14.25 (7.01)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 13.33 (5.42) | 11.44 (3.67) | 12.51 (4.75)
Weight [Mean (Standard Deviation); unit: lbs] | 191.71 (50.73) | 191.43 (47.97) | 191.57 (49.26)
Total kcals [Mean (Standard Deviation); unit: kcals] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  kcals
    Main Study Participants | 2304.47 (1022.95) | 2319.30 (781.62) | 2311.97 (907.43)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 2596.66 (1261.55) | 2506.78 (779.87) | 2563.79 (1072.38)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) is a measure of body fat based on height and weight. It is derived by dividing weight by height squared (kg/m2). Below 18.5 is underweight, 18.5 - 24.9 is a healthy weight, 25.0 - 29.9 is Overweight, and 30.0 and above is obesity.
  kg/m^2 | 29.53 (7.38) | 29.35 (6.92) | 29.44 (7.13)
Nicotine dependence [Mean (Standard Deviation); unit: units on a scale] — Fagerstrom Test for Nicotine Dependence. The Fagerstrom Test for Nicotine Dependence (FTND) is a 6-item measure with good internal consistency (α = .64) and high test-retest reliability (r = .88). Scores range from 0-8 with higher scores indicating greater nicotine dependence. The range for the SC group and the BAS group was 0-8. Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  units on a scale
    Main Study Participants | 4.75 (1.97) | 4.97 (1.79) | 4.86 (1.88)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 4.12 (1.92) | 4.68 (1.92) | 4.36 (2.40)
Substitute reinforcers [Mean (Standard Deviation); unit: Score on a scale] — Substitute reinforcers were measured by the adapted Pleasant Events Schedule, designed to assess reinforcers that occur in the natural environment. Each participant rated the 78 events once in terms of frequency (0 = none to 2 = often) and once in terms of enjoyability (0 = none to 2 = very) over a specified number of days, yielding a frequency score and an enjoyability score. The cross-product is the reinforcement from the activity. Summing the cross-products, higher scores indicated greater substitute reinforcers. Scores ranged from 0 to 165 (all), 0 to 118 (BAS), and 0 to 165 (SC). Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  Score on a scale
    Main Study Participants | 41.31 (27.25) | 40.43 (32.80) | 40.86 (30.14)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 39.68 (30.82) | 55.53 (42.33) | 46.57 (35.80)
Weight concerns [Mean (Standard Deviation); unit: score on a scale] — Weight concerns associated with quitting smoking. These concerns were measured with a reliable (α=.87) and valid 6-item scale. The items were averaged for a total score (1=not at all to 10= very much), with higher scores indicating greater concerns. The range was 1-10 (all), 1.17-10 (SC), and 1-10 (BAS). Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  score on a scale
    Main Study Participants | 4.72 (2.24) | 4.98 (2.13) | 4.85 (2.18)
    Sub-Study Participants: number analyzed (Participants) | 25 | 19 | 44
    Sub-Study Participants | 4.70 (2.07) | 4.70 (2.2) | 4.70 (2.10)
Depression Symptoms: Sub-Study [Mean (Standard Deviation); unit: units on a scale] — The 20-item Center for Epidemiologic Studies Depression Scale was used to measure depression symptoms. Likert-style response options range from 0 to 3, with a potential score range of 0 to 60. Higher scores indicate greater depression symptoms. Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  units on a scale
    number analyzed (Participants) | 25 | 19 | 44
    (all) | 11.40 (9.12) | 13.74 (7.96) | 12.41 (8.58)
Relative Reinforcement: Sub Study [Mean (Standard Deviation); unit: trials] — Participants chose between a low-effort $ reward and either a food or a $ reward of higher value and effort. Each trial presented a choice between a standard reward (27 button clicks for $0.25) or exerting greater effort to earn a higher value food or $ reward. There were 50 trials for each $ and food (participants could work 0-50 trials for either food or $), with a greater number of trials for food indicative of a higher reinforcing value of food. Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  trials
    number analyzed (Participants) | 25 | 19 | 44
    (all) | 6.19 (11.71) | 13.4 (19.3) | 9.34 (15.95)
Complementary Reinforcers: Sub-Study [Mean (Standard Deviation); unit: units on a scale] — Complementary reinforcers (CRs) were measured by the adapted Pleasant Events Schedule, assessing reinforcers in the natural environment. These are reinforcers associated with smoking. The 78 events were rated once in frequency (0=none to 2=often) and once in enjoyability (0=none to 2=very), yielding frequency and enjoyability scores. The cross-product of enjoyability x frequency were summed, with higher scores indicating greater CRs. The possible range was 0-312. Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  units on a scale
    number analyzed (Participants) | 25 | 19 | 44
    (all) | 54.20 (28.17) | 31.53 (31.15) | 44.39 (29.16)
Disinhibition: Sub-Study [Mean (Standard Deviation); unit: units on a scale] — Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
  units on a scale
    number analyzed (Participants) | 25 | 19 | 44
    (all) | 8.96 (3.45) | 10.79 (4.14) | 9.75 (3.78)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Cessation
Description: Smoking abstinence (primary outcome) will be assessed and biochemically verified at the End of Treatment Visit (week 8), at 12 and 26 weeks after the target quit date. The primary smoking outcome variable will be 7-day point prevalence abstinence (no smoking, not even a puff, for at least 7 days prior to the assessment) biochemically verified by CO < 5 ppm at End of Treatment (week 8), and by saliva cotinine < 15ng/ml at the 12- and 26-week follow-up.
Time Frame: Through Study Completion (End of Treatment Visit, 12-Week Follow-Up Visit, and 26-Week Follow-Up Visit)
Measure: Count of Participants; unit: Participants
Groups:
- Standard Counseling: Participants will attend 8 counseling sessions and receive standard smoking cessation counseling (SC).
  SC: Overeating and weight gain are common concerns reported during smoking cessation treatment. Per convention, SC will address these concerns through standard recommendations to consume low-calorie snack foods, drink water, eat nutritious meals, and exercise, but will not include skills to shape the use of these suggestions.
- Behavioral Activation: Participants will attend 8 counseling sessions and receive a behavioral activation intervention to smoking cessation and to post-cessation weight gain (BAS+).
  BAS+: The goal of the BAS+ is to maintain a level of overall reward after cessation by structuring and enhancing opportunities for reinforcement to: (1) ensure that not smoking is as reinforcing as smoking; and (2) prevent an over-reliance on food as a substitute reinforcer for smoking so that PCWG does not precipitate smoking relapse.
Arm/Group | Standard Counseling | Behavioral Activation
Number analyzed (Participants) | 146 | 142
Participants | 25 | 33

2. Primary Outcome: Weight Change
Description: Weight will be measured by a physician's scale (pounds) at the beginning of every in-person visit through study completion. Participants will be wearing light clothing without shoes. Pre-cessation weight will be computed as the average of weights at the Intake and Baseline Visits prior to any change in smoking behavior. Weight change from Baseline to the 26-week follow-up will serve as a primary weight outcome variable.
Time Frame: Through Study Completion (Intake Visit, Baseline Visit, Pre-Quit Visit , Target Quit Date Visit, Mid-Tx. 1 Visit, Mid-Tx 2 Visit, Mid-Tx 3 Visit, Mid-Tx 4 Visit , End of Treatment, 12-Week Follow-Up Visit, and 26-Week Follow-Up Visit)
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Standard Counseling | Behavioral Activation
Number analyzed (Participants) | 146 | 142
Pounds | 2.71 (12.46) | 2.00 (10.64)

3. Primary Outcome: Sub-Study: Seven-day Point Prevalence Abstinence (Carbon Monoxide) at 12 Weeks Post Target Quit Date
Description: Smoking abstinence was assessed and biochemically verified at the 12-week Follow-Up Visit (12 weeks post target quit date). Seven-day point prevalence abstinence (no smoking, not even a puff for the last 7 days prior to the assessment) was biochemically verified by a carbon monoxide (CO) reading <8 parts per million.
Time Frame: 12-Week Follow-Up Visit
Population: Sub-study: Main study participants that meet certain MRI related study criteria may also elect to complete a series of computer tasks inside a standard, closed MRI scanner to examine changes in brain activity associated with the smoking cessation counseling that participants receive in the main study. They will be asked to complete 2, one-hour fMRI scans: 1 before completing their first counseling session and 1 during the final 7 days of the scheduled 8-week nicotine patch treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Counseling: As part of the main study, participants will attend 8 counseling sessions and receive standard smoking cessation counseling (SC).
  SC: Overeating and weight gain are common concerns reported during smoking cessation treatment. Per convention, SC will address these concerns through standard recommendations to consume low-calorie snack foods, drink water, eat nutritious meals, and exercise, but will not include skills to shape the use of these suggestions.
- Behavioral Activation: As part of the main study, participants will attend 8 counseling sessions and receive a behavioral activation intervention to smoking cessation and to post-cessation weight gain (BAS+).
  BAS+: The goal of the BAS+ is to maintain a level of overall reward after cessation by structuring and enhancing opportunities for reinforcement to: (1) ensure that not smoking is as reinforcing as smoking; and (2) prevent an over-reliance on food as a substitute reinforcer for smoking so that PCWG does not precipitate smoking relapse.
Arm/Group | Standard Counseling | Behavioral Activation
Number analyzed (Participants) | 19 | 25
Participants | 9 | 10

4. Secondary Outcome: Food Intake
Description: Food intake (secondary outcome) will be assessed via 3 telephone-administered, 24-hour dietary recalls during the week after (or near) the Baseline Visit, Mid-Treatment 3 Visit (week 4), End of Treatment Visit (week 8) and the 12-week and 26-week follow-up Visits (n=15). A trained member of the research staff will use a multi-pass method with an interactive computerized software program, the Automated Self-Administered 24-hour Recall (ASA24®), to determine total kcal/day (outcome variable).
Time Frame: Through Study Completion (Baseline Visit, Mid-Tx 3 Visit, End of Treatment Visit, 12-Week Follow-Up Visit, and 26-Week Follow-Up Visit)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kcals/day
Arm/Group | Standard Counseling | Behavioral Activation
Number analyzed (Participants) | 146 | 142
kcals/day
  Main Study Participants | -156.3 (769.44) | -128.2 (943.62)
  Sub-Study Participants: number analyzed (Participants) | 19 | 25
  Sub-Study Participants | -201.85 (553.74) | 121.78 (1322.42)

5. Secondary Outcome: Sub-Study: fMRI BOLD Signal Change
Description: T2*-weighted Blood Oxygen-Level-Dependent (BOLD) images will be acquired using a wholebrain, single-shot gradient-echo (GE) echo-planar imaging (EPI) sequence. BOLD images were captured (and subsequently analyzed) while participants complete a Food Cue-Induced Craving, Relative Reinforcing Value of Food, and Working Memory task inside the MRI Scanner.
Time Frame: Pre-Treatment fMRI Scan (~week 2), End of Treatment MRI Scan (~week 8)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of signal change
Arm/Group | Standard Counseling | Behavioral Activation
Number analyzed (Participants) | 19 | 25
percentage of signal change | 0.3318 (0.22944) | -0.0003 (0.2230)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious Adverse Events were defined as any severe or serious medical event definitely related to study participation.
  Adverse Events were defined as any unanticipated medical event definitely related to study participation.
  Only Serious and Other Adverse events related to participating in the fMRI scans were monitored/assessed in the sub-study.
Groups:
- Sub-Study: Behavioral Activation: As part of the main study, participants will attend 8 counseling sessions and receive a behavioral activation intervention to smoking cessation and to post-cessation weight gain (BAS+).
- Sub-Study: Standard Counseling: As part of the main study, participants will attend 8 counseling sessions and receive standard smoking cessation counseling (SC).
Arm/Group | Behavioral Activation | Standard Counseling | Sub-Study: Behavioral Activation | Sub-Study: Standard Counseling
All-Cause Mortality (participants affected / at risk) | 0/142 | 0/146 | 0/31 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/146 | 0/31 | 0/28
Other Adverse Events (participants affected / at risk) | 0/142 | 0/146 | 0/31 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Full Study and Sub-Study (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02906787/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT02906787/ICF_001.pdf